CLINICAL TRIAL: NCT02622126
Title: The Effects of Colloid Pre-Loading on D-Dimer of the Mother and Her Baby During Cesarean Section Under Spinal Anesthesia for Mild Preeclampsia
Brief Title: Colloid Pre-Loading on D-Dimer During Cesarean Section Under Spinal Anesthesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sayed Kaoud Abd-Elshafy, Associate Professor (Anesthesiology and Critical Care)- College of Medicine-Assiut University, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB0000871175
Record Dates: First submitted 2015-12-01; First posted 2015-12-04 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Coagulation Defect; Bleeding
Keywords: Preloading; Colloid; Cesarean section; D-dimer; Hypotension
MeSH Terms: conditions — Hemostatic Disorders; Hemorrhage; Hypotension | interventions — Hydroxyethyl Starch Derivatives; HES 130-0.4; Bupivacaine; Morphine; Solutions; Saline Solution; Ephedrine; Atropine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normotensive pregnant women group (Active Comparator): Preloaded prior to spinal anesthesia with 500 mL hydroxyethyl starch (6% 130/0.4) (Voluven).
  Sub arachnoid 10-12 mg hyperbaric bupivacaine Sub arachnoid 200 meg morphine Isotonic 0.9 sodium chloride (NaCl) solution ( 10 ml/kg) will be used as co loading during the duration of the operation Ephedrine 6 me intravenous will be used to treat severe hypotension (fall of > 20% of mean arterial pressure from baseline) Atropine 0.5 mg intravenous will be used to treat bradycardia (fall of >30% of heart rate from baseline or <50 beats /minute and when associated with hypotension)
  Interventions: Drug: hydroxyethyl starch (6% 130/0.4); Drug: Hyperbaric bupivacaine; Drug: Morphine; Drug: Isotonic 0.9 sodium chloride (NaCl) solution; Drug: Ephedrine; Drug: Atropine
- Mild preeclampsia pregnant women group (Active Comparator): Preloaded prior to spinal anesthesia with 500 mL hydroxyethyl starch (6% 130/0.4) (Voluven).
  Sub arachnoid 10-12 mg hyperbaric bupivacaine Sub arachnoid 200 meg morphine Isotonic 0.9 sodium chloride (NaCl) solution (NaCl) solution ( 10 ml/kg) will be used as co loading during the duration of the operation Ephedrine 6 me intravenous will be used to treat severe hypotension (fall of > 20% of mean arterial pressure from baseline) Atropine 0.5 mg intravenous will be used to treat bradycardia (fall of >30% of heart rate from baseline or <50 beats /minute and when associated with hypotension)
  Interventions: Drug: hydroxyethyl starch (6% 130/0.4); Drug: Hyperbaric bupivacaine; Drug: Morphine; Drug: Isotonic 0.9 sodium chloride (NaCl) solution; Drug: Ephedrine; Drug: Atropine

INTERVENTIONS:
Drug: hydroxyethyl starch (6% 130/0.4) — preloaded prior to spinal anesthesia with 500 mL hydroxyethyl starch (6%130/0.4) (Voluven).
  Other Names: Voluven
Drug: Hyperbaric bupivacaine — Sub arachnoid 10-12 mg hyperbaric bupivacaine
  Other Names: Marcaine
Drug: Morphine — Sub arachnoid 200 meg morphine
Drug: Isotonic 0.9 sodium chloride (NaCl) solution — 10 ml/kg of isotonic 0.9 sodium chloride (NaCl) solutions will be used as co loading during the duration of the operation
  Other Names: Normal saline
Drug: Ephedrine — If severe hypotension (fall of > 20% of mean arterial pressure from baseline) occurred, vasopressors, 6 mg ephedrine (per dose) will be used.
Drug: Atropine — Bradycardia (fall of >30% of heart rate from baseline or <50 beats /minute and when associated with hypotension) will treated with 0.5 mg of atropine intravenous.

SUMMARY:
Maternal hypotension is the most frequent complication of a spinal Anesthesia. The prevention of spinal hypotension appears more likely to decrease the frequency and severity of associated adverse maternal symptoms than the treatment of established hypotension. Intravenous fluid administration prior to spinal anesthesia for caesarean section is accepted standard practice. The choice of fluid depends on individual and institutional habit, material cost (crystalloid is considerably cheaper) and the perceived relative benefits and risks. Uncommon but potentially serious adverse effect of colloids is impaired coagulation. Although pregnancy is associated with hypercoagulability, little is known about the effects of colloid preloading on coagulation in pregnant patients.

DETAILED DESCRIPTION:
The patients were divided into two equal group of thirty patients in each group; Control group (normotensive pregnant women) and Mild preeclampsia group. In both groups patients preloaded with 500 mL hydroxyethyl starch (HES) 6% (130/0.4) (Voluven). Spinal anesthesia will be performed with intrathecal 10-12 mg hyperbaric bupivacaine in addition to 200 meg morphine. The patient was placed supine with left lateral tilt to alleviate aortocaval compression. 10 ml/kg of isotonic 0.9 sodium chloride (NaCl) solutions will be used co loading during the duration of the operation. Blood pressure was measured and recorded every three minutes. If severe hypotension (fall of > 20% of mean arterial pressure from baseline) occurred, vasopressors, 6 mg ephedrine (per dose) will be used. The blood pressure will rechecked 1 minute after each doses of ephedrine. If hypotension persisted after 30 mg of ephedrine, an additional 2 ml/kg of isotonic 0.9 NaCl solutions will be infused rapidly. Maternal hypotension is defined as at least a single administration of ephedrine within the period from induction of spinal anesthesia until transfer to postoperative recovery unit. Reactive hypertension is characterized as a blood pressure 20% greater than baseline mean levels after the use of the vasopressor. Bradycardia is defined as a fall of >30% of heart rate from baseline or <50 beats /minute. Bradycardia, and when associated with hypotension it will be treated with 0.5 mg of atropine intravenous. Upon completion of the cesarean section, the subject will be transported to the postanesthesia care unit (PACU).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist (ASA) status I or II
* Aged >18 years
* Singleton pregnancy
* Gestational age ≥ 37 weeks
* Height ≥ 150 cm and ≤ 180 cm
* Weight > 50 kg and < 100 kg
* Eligible for spinal anesthesia
* Elective cesarean delivery

Exclusion Criteria:

* Multiple pregnancies
* Cardiovascular disease cerebrovascular disease
* Diabetes Mellitus
* Hematological problems
* Abnormal coagulation tests
* Anticoagulant use
* Hemorrhagic syndromes of pregnancy (placenta previa or accidental hemorrhage)
* Regular NSAIDS treatment
* HELLP syndrome
* Severe preeclampsia
* Eclampsia
* Termination of pregnancy for any cause
* Peripheral neuropathy or chronic pain syndrome
* Local infection or injury at the needle entry point
* Known hypersensitivity reaction to local anesthetic, starch allergy
* Height < 150 cm and > 180 cm
* Weight < 50 kg and > 100 kg
* Patient refusing spinal anesthesia
* Fetal anomalies
* Fetal distress or cases with umbilical cord prolapsed

Ages: 19 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Coagulation defect (detection of D-Dimer) of the mother | Pre and post cesarean delivery, an expected average of 90 minutes
  Blood samples for detection of D-Dimer were taken from the mother preoperatively (before colloid administration) and another one at the end of the operation
Coagulation defect (detection of D-Dimer) of the baby | Pre and post cesarean delivery, an expected average of 90 minutes
  Blood sample for detection of D-Dimer was taken from the umbilical cord of the fetus before clamping

SECONDARY OUTCOMES:
Maternal hypotension (fall of > 20% of MAP (mm Hg ) from baseline) | Post spinal for cesarean delivery, an expected average of 4 hours
  fall of > 20% of MAP (mm Hg ) from baseline
Ephedrine treatment (Ephedrine total dosage (mg)) | Post spinal for cesarean delivery, an expected average of 4 hours
  Ephedrine total dosage (mg)
Atropine treatment (atropine total dosage (mg)) | Post spinal for cesarean delivery, an expected average of 4 hours
  atropine total dosage (mg)
Hemoglobin concentration | Pre and post cesarean delivery, an expected average of 4 hours
  Blood samples for detection of hemoglobin concentration gm/dL
Platelet count | Pre and post cesarean delivery, an expected average of 4 hours
  Blood samples for detection of platelet count (109/L )

CONTACTS AND LOCATIONS:
Overall Officials: sayed abd elshafy, MD, Principal Investigator — associate professor
Locations (1):
- Faculty of Medicine, Asyut, Asyut Governorate, Egypt